CLINICAL TRIAL: NCT00765271
Title: A Study Investigating Plasma Abacavir and Its Intracellular Anabolite Carbovir-triphosphate Pharmacokinetics in the Absence and in the Presence of Darunavir/Ritonavir or Raltegravir in HIV-infected Subjects.
Brief Title: Abacavir Pharmacokinetic Study in the Absence/Presence of Darunavir/Ritonavir or Raltegravir in HIV-infected Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St Stephens Aids Trust (Other)
Responsible Party: Dr Marta Boffito, St Stephen's AIDS Trust
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SSAT026; EudraCT No: 2007-005965-37 (Other: EU Clinical Trials Database)
Record Dates: First submitted 2008-10-01; First posted 2008-10-02 (Estimated); Last update posted 2009-11-18 (Estimated); Status verified 2009-11

CONDITIONS: HIV
MeSH Terms: interventions — abacavir; abacavir, lamivudine, and zidovudine drug combination; abacavir, lamivudine drug combination; Darunavir; Ritonavir; Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 2 (Active Comparator): Abacavir 600 mg (2 x 300mg tablet) once daily throughout the study (days 1- 30) Raltegravir 400 mg (2 x 200mg tablets) twice daily from days 2 to 15 Darunavir/ritonavir 900 (3 x 300mg tablets)/100 (1 x 100mg capsule) mg once daily from day 16 to day 29)
  Interventions: Drug: Abacavir; Drug: Raltegravir
- Group 1 (Active Comparator): Abacavir 600 mg (2 x 300mg tablet) once daily throughout the study (days 1- 30) Darunavir/ritonavir 900 (3 x 300mg tablets)/100 (1 x 100mg capsule) mg once daily from day 2 to day 15) Raltegravir 400 mg (2 x 200mg tablets) twice daily from day 16 to 29
  Interventions: Drug: Abacavir; Drug: Darunavir/ritonavir; Drug: Raltegravir

INTERVENTIONS:
Drug: Abacavir — Group 1 will be instructed to take • Abacavir 600 mg once daily (two 300 mg tablets once daily) as part of regular treatment throughout the whole study
  Group 2 will be instructed to take
  • Abacavir 600 mg once daily (two 300 mg tablets once daily) as part of regular treatment throughout the whole study
  Other Names: Ziagen®; Trizivir®; Kivexa®.
Drug: Darunavir/ritonavir — Group 1 will be instructed to take
  • Three 300mg Darunavir tablets and one 100mg ritonavir tablet once a day for 14 days (on days 2 - 15)
  Arms: Group 1
Drug: Raltegravir — Group 1 will be instructed to take • Two 200mg Raltegravir tablets twice daily for 14 days (on 16 - 29)
  Group 2 will be instructed to take
  • Two 200mg Raltegravir tablets twice daily for 14 days (on days 2-15)

SUMMARY:
The study is being conducted as we have found that many patients with Human Immunodeficiency Disease (HIV) require a combination of different drugs to treat the HIV infection. Before using different combination of drugs, it is important to do studies to see if the drugs will affect the activity of one another.

The study aims to help us understand if darunavir/ritonavir or raltegravir have any effects on levels of abacavir in the blood.

The purpose of the study is to assess the pharmacokinetics (how a drug is absorbed, distributed and eliminated from your body) of abacavir in the absence and in the presence of darunavir/ritonavir and raltegravir.

DETAILED DESCRIPTION:
Since the co-administration of nucleoside analogues and protease inhibitors, and soon integrase inhibitors, forms an integral part of highly active antiretroviral therapy (HAART) and these combinations may result in unexpected drug interactions (as demonstrated by interactions between protease inhibitors and TFV), it is therefore important to elucidate the impact of ARV co-administration on drug levels.

The risk of ABC hypersensitivity (HSR) precludes the study of this agent in healthy volunteers therefore this study will be performed in HIV-infected subjects. Clinical efficacy of drugs is related to their plasma concentrations [Boffito, 2005] and it is important to know whether ABC has any impact on the levels of therapeutic agents that may impact on their clinical efficacy. Moreover, it is still unknown whether ABC exposure is altered by the ritonavir-boosted protease inhibitors darunavir or by the new HIV drug raltegravir. Raltegravir will be soon approved for the treatment of HIV in Europe and United States.

Pharmacogenetics holds promise in HIV treatment because of the complexity and potential toxicity of multi antiretroviral drug therapies that are prescribed for long periods. Thus far, few candidate genes have been examined for a limited number of allelic variants, but a number of confirmed associations have already emerged.

From a public health perspective, as antiretroviral medications become increasingly available to racially and ethnically diverse populations worldwide, understanding the genetic structures of each population may allow us to anticipate the impact of adverse responses, even in groups that were not represented in drug registration trials.

The existing literature on pharmacogenetic determinants of antiretroviral drug exposure, drug toxicity, as well as genetic markers associated with the rate of disease progression underline the recent advances which occurred in the past few years.

However, it is expected that larger-scale comprehensive genome approaches will profoundly change the landscape of knowledge in the future. Additional studies are needed to assess the implications for long-term responses to antiretroviral agents.

For this reason we plan to collect a single blood sample from each participant in our intensive pharmacokinetic studies, such as this one, in order to be able to investigate the association between genetic polymorphisms in drug disposition genes (such as those encoding for cytochrome P450 isoenzymes or transmembrane transporters) and drug exposure. A candidate gene approach will be utilised to examine loci of interest. This procedure will provide potentially important information on genetic influences on plasma drug concentrations and give insight into how to improve the management of HIV-infected patients by individualising therapy. These studies will not be powered for genetic associations but will enable us to build a data base of genotype-phenotype. Prospective genetic studies would need to be planned based on these preliminary data.

ELIGIBILITY:
Inclusion Criteria:

1. The ability to understand and sign a written informed consent form, prior to participation in any screening procedure and must be willing to comply with all study requirements.
2. Male or non-pregnant, non-lactating females.
3. Between 18 to 65 years, inclusive.
4. Documented HIV-1 infection and plasma HIV RNA at screening visit below 400 copies/mL. (Note retesting of screening viral load is allowed).
5. CD4 count > 100 at screening (Note retesting of screening CD4 count is allowed).
6. Receiving an abacavir-containing regimen which does not include tenofovir, a protease inhibitor, a non-nucleoside reverse transcriptase inhibitor or a fusion inhibitor at screening.
7. Agrees not to change regimen from baseline until end of the treatment period unless this is medically indicated as decided by the treating physician.

Exclusion Criteria:

1. Any serious or active medical or psychiatric illness which, in the opinion of the investigator, would interfere with subject treatment, assessment, or compliance with the protocol. This would include any active clinically significant renal, cardiac, hepatic, pulmonary, vascular, metabolic disorders or malignancy.
2. Have a body mass index (BMI) >30
3. Presence of any current active AIDS defining illness (Category C conditions according to the CDC Classification System for HIV Infection 1993) with the following exceptions:

   • Stable cutaneous Kaposi's Sarcoma
4. Clinically relevant alcohol or drug use (positive urine drug screen) or history of alcohol or drug use considered by the Investigator to be sufficient to hinder compliance with treatment, follow-up procedures or evaluation of adverse events. Smoking is permitted, but tobacco intake should remain consistent throughout the study.
5. Concurrent use of non-nucleoside reverse transcriptase inhibitors (NNRTIs), protease inhibitors, fusion inhibitors or tenofovir.

7. The use of disallowed concomitant therapy (See Concomitant Medication and treatment, section 5.2).

8. Females of childbearing potential without the use of effective non-hormonal birth control methods or not willing to continue practicing these birth control methods for at least 14 days after the end of the treatment period.

9. Previous allergy to any of the constituents of the pharmaceuticals administered in this trial.

10. Subjects with clinical or laboratory evidence of significantly decreased hepatic or renal function (as determined by the principal investigator).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2008-05; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Steady state plasma concentrations of abacavir and intracellular concentrations of its active anabolite carbovir-TP following the administration of abacavir 600 mg once daily, in the absence and in the presence of darunavir/ritonavir or raltegravir | 30 days

SECONDARY OUTCOMES:
Plasma pharmacokinetics of darunavir/ritonavir and raltegravir in the presence of abacavir in HIV-infected subjects Safety and tolerability of abacavir in the presence of darunavir/ritonavir or raltegravir in HIV-infected subjects | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Marta Boffito, Principal Investigator — St Stephen's AIDS Trust
Locations (1):
- Chelsea and Westminster Hospital, London, London, United Kingdom